CLINICAL TRIAL: NCT00543426
Title: Fuzheng Huayu Tablets Against Posthepatitic Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06DZ19728
Record Dates: First submitted 2007-10-12; First posted 2007-10-15 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2009-06

CONDITIONS: Posthepatitic Cirrhosis
Keywords: Fuzheng Huayu Tablets; Multicenter clinical study
MeSH Terms: interventions — fuzheng huayu

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Fuzheng Huayu Tablets
  Interventions: Drug: Fuzheng Huayu Tablets
- 2 (Sham Comparator): sham Fuzheng Huayu Tablets
  Interventions: Drug: sham Fuzheng Huayu Tablets (placebo)

INTERVENTIONS:
Drug: Fuzheng Huayu Tablets — Tablet,three times a day,four tablets one time
  Arms: 1
Drug: sham Fuzheng Huayu Tablets (placebo) — Tablet, three times a day, four tablets one time
  Arms: 2

SUMMARY:
The primary purpose of the trial is adopted Fuzheng Huayu tablets against posthepatitic cirrhosis, and to build a standard evaluation system for efficacy of traditional Chinese medicine (TCM).

The second purpose is according to the international clinical guideline and the specialty of TCM to build a standard clinical trial regulation for traditional Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of B Post hepatitic cirrhosis.
* Male or female patients between 18~65 years old.
* Written informed consent.

Exclusion Criteria:

* Child-Pugh C above 12, or ALT > 2×ULN, TBiL > 2×ULN, or combined with hepatic encephacopathy, Obstinate ascites, bleeding tendency, hepato-renal syndrome, or primary liver cancer.
* Combined with severe heart, gallbladder, kidney, endocrine system, hemopoietic system or nervous system disease.
* Deformed man by the law.
* Pregnancy or breast feeding women, or unwilling to have contraception.
* Irritability body constitution, or irritability of the Fuzheng Huayu Capsules.
* Enter other trials lately one month.
* Other cause of cirrhosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-09; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
the value of Child-Pugh and symptoms scale for Posthepatitic Cirrhosis | six months

SECONDARY OUTCOMES:
hepatic function; blood test; blood ammonia and blood sugar determination | six months

CONTACTS AND LOCATIONS:
Overall Officials: Zengzeng Cai, Ph.D, Study Director — Shanghai Univercity of TCM
Locations (1):
- Shuguang Hospital, Shanghai, China

REFERENCES:
- [Background] Zhao CQ, Wu YQ, Xu LM. [Curative effects of Fuzheng Huayu capsules on hepatic fibrosis and the functional mechanisms: a review]. Zhong Xi Yi Jie He Xue Bao. 2006 Sep;4(5):467-72. doi: 10.3736/jcim20060505. Chinese. PMID 16965738
- [Background] Liu P, Hu YY, Liu C, Xu LM, Liu CH, Sun KW, Hu DC, Yin YK, Zhou XQ, Wan MB, Cai X, Zhang ZQ, Ye J, Tang BZ, He J. [Multicenter clinical study about the action of Fuzheng Huayu Capsule against liver fibrosis with chronic hepatitis B]. Zhong Xi Yi Jie He Xue Bao. 2003 Jul;1(2):89-98, 102. doi: 10.3736/jcim20030204. Chinese. PMID 15339577
- [Background] Zhang Q, Zhang WT, Wei JJ, Wang XB, Liu P. [Combined use of factor analysis and cluster analysis in classification of traditional Chinese medical syndromes in patients with posthepatitic cirrhosis]. Zhong Xi Yi Jie He Xue Bao. 2005 Jan;3(1):14-8. doi: 10.3736/jcim20050105. Chinese. PMID 15644152